CLINICAL TRIAL: NCT04735978
Title: An Open-Label, Multicenter, Phase 1 Study of RP3 as a Single Agent and in Combination With PD-1 Blockade in Patients With Solid Tumors
Brief Title: Study of RP3 Monotherapy and RP3 in Combination With Nivolumab in Patients With Solid Tumours
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Replimune Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RP3-301
Record Dates: First submitted 2021-01-25; First posted 2021-02-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced solid tumors; Immunotherapy; Immuno-oncology; Oncolytic virus; Oncolytic immuno-gene therapy
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Part 1 - Dose Escalation - Participants will be enrolled into two sequential dose level cohorts.
  * Cohort 1: 1 × 105 plaque-forming units (PFU)/mL on Day 1 followed by 1 × 106 PFU/mL every 2 weeks (Q2W) for up to 5 doses.
  * Cohort 2: 1 × 106 PFU/mL on Day 1 followed by 1 × 107 PFU/mL Q2W for up to 5 doses.
  Part 2 - Dose Combination - Patients will be enrolled into 1 of 5 dose-expansion cohorts. Expansion Cohorts 1, 2, and 4 will enroll patients with head and neck cancer, lung cancer, breast cancer, or GI cancer. Expansion Cohort 3 will enroll patients with any solid organ malignancy who have at least 2 tumors that can be injected and biopsied. Expansion Cohort 5 will enroll patients with melanoma.
  * Expansion Cohort 1 (RP3 + Nivolumab)
  * Expansion Cohort 2 (RP3 Followed by Nivolumab)
  * Expansion Cohort 3 (RP3 Monotherapy Translational Cohort)
  * Expansion Cohort 4 (RP3 Monotherapy)
  * Expansion Cohort 5 (RP3 + Nivolumab in Melanoma)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose escalation of RP3 - superficial and/or deep/visceral tumors (Experimental): Dose escalation of RP3 alone in 2 cohorts with intratumoral (IT) injections including use of imaging guided injection for deep tumors.
  Interventions: Biological: RP3
- Dose combination of RP3 and anti-PD1 therapy - superficial and/or deep/visceral tumors (Experimental): Dose combination of RP3 and anti-PD1 therapy. IT injections of RP3 including use of imaging guided injection for deep tumors.
  Interventions: Biological: RP3; Biological: Nivolumab
- Seronegative cohort (Experimental): Doses of RP3 (IT) in HSV seronegative participants.
  Interventions: Biological: RP3

INTERVENTIONS:
Biological: RP3 — Genetically modified HSV-1
Biological: Nivolumab — anti-PD1 monoclonal antibody
  Arms: Dose combination of RP3 and anti-PD1 therapy - superficial and/or deep/visceral tumors

SUMMARY:
This is a Phase 1, multicenter, open label, single agent dose escalation and combination treatment study of RP3 in adult participants with advanced solid tumors, to evaluate the safety and tolerability of RP3 both as a single agent and in combination with anti-PD1 therapy and to determine the recommended Phase 2 dose (RP2D) of RP3.

DETAILED DESCRIPTION:
RP3 is a genetically modified herpes simplex type 1 virus (HSV-1) that expresses exogenous genes (anti-CTLA-4 antibody, CD40 ligand and h4-1BBL) designed to directly destroy tumors and generate an anti-tumor immune response

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic non-neurological solid tumors, who have progressed on standard therapy or cannot tolerate standard therapy, or for whom there is no standard therapy preferred to enrollment in a clinical study
* All patients must consent to provide archival tumor biopsy samples within 12 months, or a fresh tumor biopsy is needed. Patients must also consent to provide on treatment biopsies as per protocol
* At least one measurable tumor ≥ 1 cm in longest diameter (or shortest diameter for lymph nodes)
* At least one injectable tumor ≥ 1 cm in longest diameter or injectable tumors which in aggregate are ≥ 1 cm in longest diameter (or shortest diameter for lymph nodes
* Have an Eastern Cooperative Oncology Group (ECOG) performance status 0-1

Note: Predefined inclusion criteria may apply for each additional expansion cohort.

Exclusion Criteria:

* Prior treatment with an oncolytic virus therapy
* History of viral infections according to the protocol
* Systemic infection requiring intravenous (IV) antibiotics
* Active significant herpetic infections or prior complications of HSV-1 infection (e.g., herpetic keratitis or encephalitis)
* Requires intermittent or chronic use of systemic antivirals

  a. Hepatocellular carcinoma patients with a diagnosis of hepatitis B must be off antiviral therapy for at least 4 weeks prior to enrollment . Hepatocellular carcinoma patients with a history of or ongoing hepatitis C infection must have completed treatment for hepatitis C at least 1 month prior to study enrollment and hepatitis
* History of interstitial lung disease
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis

Additional Exclusion Criteria for Patients Enrolled in Part 2 (Expansion Cohorts):

* History of life-threatening toxicity related to prior immune treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Treatment with botanical preparations within 2 weeks prior to treatment.
* Active, known, or suspected autoimmune disease requiring systemic treatment.
* History of interstitial lung disease.
* Severe hypersensitivity to another monoclonal antibody.
* Has received prior radiotherapy within 2 weeks of start of study treatment.
* Has received a live vaccine within 28 days prior to the first dose of study treatment.
* History of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* History of myocarditis or congestive heart failure within 6 months of screening.
* Has a serious or uncontrolled medical disorder.
* Has a QT interval corrected for heart rate using Fridericia's formula (QTcF) > 480 msec, except for right bundle branch block.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2020-12-29 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) during the DLT period | From Day 1 up to 30 days after last dose
  Percentage of participants with DLTs
Incidence and severity of treatment emergent adverse events (TEAEs) | From Day 1 up to 60 days after last dose
  Percentage of participants with TEAEs
Incidence and severity of serious adverse events (SAEs) | From Day 1 up to 60 days after last dose
  Percentage of participants with SAEs
Incidence of TEAEs ≥ Grade 3 | From Day 1 up to 60 days after last dose
  Percentage of participants with TEAEs ≥ Grade 3
Percentage of events requiring withdrawal | From Day 1 up to last dose (up to 8 weeks in escalation phase and up to 2 years in combination phase)
  Percentage of participants experiencing events requiring withdrawal from treatment.
Recommended phase 2 dose (RP2D) of RP3 | 7 months
  RP2D of RP3 based on the safety and response data collected during the dose escalation phase (Part 1)

SECONDARY OUTCOMES:
Percentage of biologic activity | From Day 1 to 24 months following the last dose in dose escalation. From Day 1 to 100 days following the last dose in dose combination
  Percentage of participants with biological activity as assessed by individual tumor responses (including erythema, necrosis, and/or inflammation and changes in tumor sizes, in injected and uninjected tumors).
Incidence of clearance of RP3 from blood and urine | From Day 1 to 60 days following the last dose in dose escalation. From Day 1 to 100 days following the last dose in dose combination
  Incidence of clearance of RP3 from blood and urine before and after each injection
Percentage of participants with detectable RP3. | From Day 1 to 60 days following the last dose in dose escalation. From Day 1 to 100 days following the last dose in dose combination
  Data gathered from blood, urine, swabs of injection site, dressing and oral mucosa to determine the shedding and biodistribution of RP3
Change in HSV-1 antibody levels | From Day 1 to Day 43
  Change in HSV-1 antibody levels during treatment compared to baseline
Percentage of HSV-1 seronegative patients with TEAEs | From Day 1 to 60 days following last dose in dose escalation. From Day 1 to 100 days post last dose in dose combination
  Percentage of HSV-1 seronegative patients with TEAEs
Percentage of objective overall response rate (ORR) | Up to 3 years since first patient in
  Percentage of ORR
Median duration of response | Up to 3 years since first patient in
  Median duration of response of participants
Percentage of complete response (CR) | From Day 1 up to last dose (Day 57 or 8th Re-initiation dose in escalation phase and up to 2 years for combination phase)
  Percentage of participants with a CR
Percentage of partial response (PR) | From Day 1 up to last dose (Day 57 or 8th Re-initiation dose in escalation phase and up to 2 years for combination phase)
  Percentage of participants with a PR
Percentage of stable disease (SD) | From Day 1 up to last dose (Day 57 or 8th Re-initiation dose in escalation phase and up to 2 years for combination phase)
  Percentage of participants with SD
Progression-free survival by Investigator review | From Day 1 to day of last follow-up
  Length of time during and after treatment, that a patient lives with disease but it does not get worse
One-year and 2-year OS rates | From Day 1 to Day 730
  Percentage of participants from Day 1 of treatment who reach one year or two year survival

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Kumar, MD, Study Director — Replimune Inc.
Locations (13):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
- Laboratoire de Recherche Translationnelle en Immunotherapie (LRTI), Gustave Roussy, Villejuif, France
- Greece (2):
  - University of Athens, Athens
  - University General Hospital Attikon, Athens
- Spain (4):
  - Vall d'Hebron Hospital Hospital Universitario Vall d´Hebron (Vall d'Hebron University Hospital), Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - START Madrid CIO Clara Campal, Hospital Universitario HM Sanchinarro Unidad de Ensayos Fase I Panta 3, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia
- United Kingdom (3):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Merseyside
  - The Royal Marsden NHS Foundation Trust, London
  - Churchill Hospital, Oxford